CLINICAL TRIAL: NCT00284297
Title: Follow-up of Patients After Knee Arthrodesis With an Intramedullary Nail
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005/213
Record Dates: First submitted 2006-01-30; First posted 2006-01-31 (Estimated); Last update posted 2022-12-20 (Actual); Status verified 2014-12

CONDITIONS: Knee Arthrodesis With Intramedullary Nail
MeSH Terms: interventions — Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- knee arthrodesis (Experimental)
  Interventions: Procedure: History taken and clinical examination

INTERVENTIONS:
Procedure: History taken and clinical examination — History is taken and clinical examination is followed

SUMMARY:
Follow-up of patients who underwent a knee arthrodesis with different types of intramedullary nails.

ELIGIBILITY:
Inclusion Criteria:

* All patients who underwent a knee arthrodesis with an intramedullary nail between 1994 and 2005

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-09 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Follow-up of patients who underwent a knee arthrodesis with different types of intramedullary nails | t0

CONTACTS AND LOCATIONS:
Overall Officials: René Verdonk, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be